CLINICAL TRIAL: NCT01836068
Title: Optimized Antiretroviral Therapy During Allogeneic Hematopoietic Stem Cell Transplantation in HIV-1-infected Individuals
Brief Title: Optimized Antiretroviral Therapy During Allogeneic Hematopoietic Stem Cell Transplantation in HIV-1 Individuals
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: J1331; NA_00083734 (Other: Johns Hopkins); 1P30AI094189-01A1 (NIH)
Record Dates: First submitted 2013-04-16; First posted 2013-04-19 (Estimated); Last update posted 2021-11-23 (Actual); Status verified 2021-06

CONDITIONS: HIV
Keywords: HIV positive; HIV-1; Bone Marrow Transplant; Allogeneic BMT; BMT
MeSH Terms: conditions — HIV Seropositivity | interventions — Enfuvirtide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enfuvirtide monotherapy (Experimental): Enfuvirtide 90 mg subcutaneously every 12 hours will be also be administered during any periods when oral medications are not expected to be tolerated for ≥ 24 hours, or during periods when ART is held due to interactions with conditioning regimens in patients who require ritonavir-boosted PI containing ART regimens.
  Interventions: Drug: Enfuvirtide

INTERVENTIONS:
Drug: Enfuvirtide — Enfuvirtide 90 mg subcutaneously twice daily will be administered to all patients on day 3 and 4 post-transplant and during any periods when oral medications are not expected to be tolerated for ≥ 24 hours, or during periods when ART is held due to interactions
  Other Names: Fuzeon

SUMMARY:
To find out if it is possible for HIV-1 patients to maintain antiretroviral medications during allogeneic bone marrow transplant

DETAILED DESCRIPTION:
Determine the feasibility of maintaining optimal ART in HIV-1 infected patients during allogeneic hematopoietic stem cell transplant (HSCT). The primary outcome is the fraction of patients who maintain any form of anti-retroviral therapy, including enfuvirtide monotherapy, through day 60 post-transplant. If patients are unable to take oral anti-retroviral medications, but are able to tolerate subcutaneous enfuvirtide monotherapy this will be considered maintenance of ART. Failure to maintain ART will be defined as ≥ 24 hours without any anti-retroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, as documented by a rapid HIV-1 test or any FDA-approved HIV-1 enzyme or chemiluminescence immunoassay (E/CIA) test kit and confirmed by western blot at any time prior to study entry. Alternatively, two HIV-1 RNA values > 200 copies/mL at least 24 hours apart performed by any laboratory that has CLIA certification, or its equivalent may be used to document infection.
* Patients must be ≥ 18 years of age.
* Plan to undergo a Myeloablative, HLA matched or partially HLA-mismatched (haploidentical), related-donor bone marrow transplantation that includes high-dose posttransplantation Cy using bone marrow from a related donor:
* Plan to undergo a Nonmyeloablative, HLA matched or partially HLA-mismatched, related-donor bone marrow transplantation that includes high-dose posttransplantation Cy using bone marrow from a related donor:

Exclusion Criteria:

* Patients with a known history of enfuvirtide resistance will not be eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2021-06-05 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility of maintaining optimal ART in HIV-1 infected patients during allogeneic HSCT | 24 hours
  Failure to maintain anti retroviral therapy for 24 hours

SECONDARY OUTCOMES:
Number of copies of HIV-1 DNA in blood mononuclear cells at baseline | Baseline
  Measure the number of copies of HIV-1 DNA per million peripheral blood mononuclear cells.
Number of copies of HIV-1 DNA in blood mononuclear cells at 12 weeks | 12 weeks post-intervention
  Measure the number of copies of HIV-1 DNA per million peripheral blood mononuclear cells.
Number of copies of HIV-1 DNA in blood mononuclear cells at 24 weeks | 24 weeks post-intervention
  Measure the number of copies of HIV-1 DNA per million peripheral blood mononuclear cells.
Number of copies of HIV-1 DNA in blood mononuclear cells at 36 weeks | 36 weeks post-intervention
  Measure the number of copies of HIV-1 DNA per million peripheral blood mononuclear cells.
Number of copies of HIV-1 DNA in blood mononuclear cells at 52 weeks | 52 weeks post-intervention
  Measure the number of copies of HIV-1 DNA per million peripheral blood mononuclear cells.
Number of copies of HIV-1 DNA in blood mononuclear cells at 2 years | 2 years post-intervention
  Measure the number of copies of HIV-1 DNA per million peripheral blood mononuclear cells.

OTHER OUTCOMES:
The incidence of acute graft-vs-host disease | 2 years post-intervention
  Describe the incidence of acute graft-vs-host disease via the Keystone criteria
The severity of acute graft-vs-host disease | 2 years post-intervention
  Describe the severity of acute graft-vs-host disease via the Keystone criteria
The incidence of chronic graft-vs-host disease as defined by the NIH consensus criteria | 2 years post-intervention
  Describe the incidence chronic graft-vs-host disease via the NIH consensus criteria.
The incidence of chronic graft-vs-host disease as defined by the Seattle criteria | 2 years post-intervention
  Describe the incidence chronic graft-vs-host disease via the Seattle criteria.
The severity of chronic graft-vs-host disease as defined by the NIH consensus criteria | 2 years post-intervention
  Describe the severity of chronic graft-vs-host disease via the NIH consensus criteria and the Seattle criteria
The severity of chronic graft-vs-host disease as defined by the Seattle criteria | 2 years post-intervention
  Describe the severity of chronic graft-vs-host disease via the Seattle criteria

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ambinder, M.D., Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Capoferri AA, Redd AD, Gocke CD, Clark LR, Quinn TC, Ambinder RF, Durand CM. Brief Report: Rebound HIV Viremia With Meningoencephalitis After Antiretroviral Therapy Interruption After Allogeneic Bone Marrow Transplant. J Acquir Immune Defic Syndr. 2022 Mar 1;89(3):297-302. doi: 10.1097/QAI.0000000000002862. PMID 34753870
- [Derived] Capoferri AA, Redd AD, Gocke CD, Clark LR, Ambinder RF, Durand CM. Short Communication: Persistence of HIV After Allogeneic Bone Marrow Transplant in a Dually Infected Individual. AIDS Res Hum Retroviruses. 2022 Jan;38(1):33-36. doi: 10.1089/AID.2021.0047. Epub 2021 Jul 5. PMID 34107771
- [Derived] Durand CM, Capoferri AA, Redd AD, Zahurak M, Rosenbloom DIS, Cash A, Avery RK, Bolanos-Meade J, Bollard CM, Bullen CK, Flexner C, Fuchs EJ, Gallant J, Gladstone DE, Gocke CD, Jones RJ, Kasamon YL, Lai J, Levis M, Luznik L, Marr KA, McHugh HL, Mehta Steinke S, Pham P, Pohlmeyer C, Pratz K, Shoham S, Wagner-Johnston N, Xu D, Siliciano JD, Quinn TC, Siliciano RF, Ambinder RF. Allogeneic bone marrow transplantation with post-transplant cyclophosphamide for patients with HIV and haematological malignancies: a feasibility study. Lancet HIV. 2020 Sep;7(9):e602-e610. doi: 10.1016/S2352-3018(20)30073-4. Epub 2020 Jul 7. PMID 32649866